CLINICAL TRIAL: NCT04280848
Title: Anticancer Therapeutic Vaccination Using Telomerase-derived Universal Cancer Peptides in Glioblastoma
Acronym: UCPVax-Glio
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N/2013/67
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: UCPVax vaccine (patient with unmethylated MGMT status) (Experimental): UCPVax
  Interventions: Drug: UCPVax
- Cohort B: UCPVax vaccine + Temozolomide (patient with unmethylated or methylated MGMT status) (Experimental): UCPVax
  + Temozolomide according to standard of care
  Interventions: Drug: UCPVax; Drug: Temozolomide

INTERVENTIONS:
Drug: UCPVax — The UCPVax vaccination protocol will start at least one month after glioblastoma patients have completed the concomitant radiochemotherapy (Radiotherapy + Temozolomide RT/TMZ).
  UCPVax vaccine will injected subcutaneously at days 1, 8, 15, 29, 36 and 43 (priming phase) following by boost vaccination one month after the last injection and then every 8 weeks for 12 months maximum.
Drug: Temozolomide — 6 additional monthly cures of Temozolomide (after concomitant radiotherapy and temozolomide) according to standard of care
  Arms: Cohort B: UCPVax vaccine + Temozolomide (patient with unmethylated or methylated MGMT status)

SUMMARY:
Glioblastoma (GBM) is the most frequent primary brain tumor and the brain tumor with the poorest prognosis. The current treatment relies on surgical resection of gross tumor followed by radiochemotherapy and adjuvant therapy with temozolomide.

After such therapy, most patients experiment recurrence and few therapeutic option are available. Despite such therapies, median survival only reaches around fifteen months.

There is a strong rational to develop telomerase vaccine in GBM. Telomerase (TERT) is a major oncogene, particularly in primary brain tumors 24. Alterations in TERT are very frequent in central nervous system tumors, seen most commonly in gliomas25. Mutations in the TERT promoter are found in approximately 80% of primary glioblastoma (GBM). These findings strongly support the rational to develop vaccine targeting telomerase in GBM.

The aim of this project is to evaluate UCPVax treatment in glioblastoma. UCPVax is a therapeutic anti-cancer vaccine based on the telomerase-derived helper peptides designed to induce strong TH1 CD4 T cell responses in cancer patients (NCT02818426).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≥ 18 and ≤ 75 years old
* Written informed consent
* Histologically confirmed glioblastoma
* Patient with known MGMT status:

Cohort A (recruitment closed) : unmethylated MGMT status ; Cohort B (recruiting) : unmethylated or methylated MGMT status

* Patients previously pre-treated with standard radiochemotherapy (without the additional cures of temozolomide.)
* Karnofsky Performance status ≥ 70%
* Life-expectancy > 3 months
* Adequate hematological, hepatic, and renal function.
* Females must be using highly effective contraceptive measures , and have a negative pregnancy test prior to the start of dosing if of childbearing potential, or must have evidence of non-childbearing potential.

Females of childbearing potential should use reliable methods of contraception from the time of the screening until 5 weeks after discontinuing study treatment.

Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 5 months following discontinuation of study drug. Patients should refrain from donating sperm from the start of dosing until 5 months after discontinuing study treatment.

- Affiliation to French social security or receiving such a regime.

Exclusion Criteria:

* Presence of known extracranial metastatic or leptomeningeal disease Glioblastoma with mutated IDH1 (assessed by Immunohistochemistry)
* Current or recent treatment with another investigational drug
* Carmustine implant during surgery
* History of autoimmune diseases (lupus, rheumatoid arthritis, inflammatory bowel disease…)
* Prohibited medications:

  1. Chronic treatment with immunosuppressive drugs
  2. Ongoing requirement for supraphysiologic steroid defined as >10 mg prednisone daily (or equivalent)
  3. Treatment with therapeutic oral or IV antibiotics within 4 weeks prior to enrollment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or pulmonary disease) are eligible for the study
* Known positive serology for Human Immunodeficiency Virus (HIV) or Hepatitis C virus (HCV); presence in the serum of the antigens HBs
* Non-hematologic toxicities Grade >1 severity (or, at the investigator's discretion, Grade >2 if not considered a safety risk for the patient).
* Patient with intra-alveolar hemorrhage, pulmonary fibrosis, or uncontrolled asthma, or chronic obstructive disease (COPD), defined as at least 1 hospitalization within 4 months prior to enrollment or as at least 3 exacerbations during the last year prior to enrollment Hospitalization for cardiovascular or pulmonary disease within 4 weeks prior to enrollment.
* Patients with LEVF<40%
* Participation in a clinical study with an investigational product within 4 weeks prior to the start of the study treatment or patient in the exclusion period of a previous clinical trial.
* Pregnancy or lactating patients.
* Patients with any severe/uncontrolled inter current illness, significant co morbid or psychiatric conditions that in the opinion of the investigator would impair study participation or cooperation.
* Patients under guardianship, curatorship or under the protection of justice.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | at day 60
  Anti-TERT specific T cell responses measured in peripheral blood using IFN-gamma ELISPOT

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde VERLUT, Dr, Principal Investigator — CHU Besançon
Locations (5):
- France (5):
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - CHU La Timone, Marseille
  - Hôpital Saint-Louis, Paris